CLINICAL TRIAL: NCT02492802
Title: Effect of Inflammation on Pharmacokinetics of Posaconazole
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jan-Willem C Alffenaar, PharmD PhD, University Medical Center Groningen
Other Study IDs: POSA-CRP
Record Dates: First submitted 2015-07-02; First posted 2015-07-09 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Mycoses
MeSH Terms: conditions — Mycoses | interventions — posaconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- posaconazole-group: patients receiving posaconazole for prophylaxis or treatment of invasive fungal infection
  Interventions: Drug: posaconazole

INTERVENTIONS:
Drug: posaconazole — collection plasma samples for measuring posaconazole drug concentration
  Other Names: noxafil

SUMMARY:
Posaconazole plasma concentration and inflammatory markers will be determined in all samples available from routine analysis.

DETAILED DESCRIPTION:
A prospective observational study will be performed at the University Medical Center Groningen, the Netherlands using longitudinal data collection. The design of the study will be that patients starting on posaconazole treatment will be evaluated. After informed consent is obtained medical data will be collected from the medical chart. Posaconazole plasma concentration (trough levels) and inflammatory markers (e.g. C-reactive protein) will be determined in all samples available from routine analysis (often daily). This will result in a detailed data set capturing day to day variations in inflammation and drug concentrations.

ELIGIBILITY:
Inclusion Criteria:

* >18 yrs
* receiving posaconazole
* Written informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * patients with hematological malignancies
  * immunocompromised patients
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem Alffenaar, PharmD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients on Posaconazole: Hematology patients receiving posaconazole for routine care.
Period: Overall Study
Arm/Group | Patients on Posaconazole
Started | 64
Completed | 64
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients on Posaconazole: Patient characteristics and drug dosing information (oral and intravenous dosing, daily dose of posaconazole)
Arm/Group | Patients on Posaconazole
Number analyzed (Participants) | 64
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [55 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 64
Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 79 [71 to 86]
Height (cm) [Median (Inter-Quartile Range); unit: cm] | 178 [171 to 184]
Acute myeloid leukemia [Count of Participants; unit: Participants] | 40
Myelodysplastic syndrome [Count of Participants; unit: Participants] | 10
Other underlying disease [Count of Participants; unit: Participants] | 14
Allogeneic stem cell transplant [Count of Participants; unit: Participants] | 22
Autologous stem cell transplant [Count of Participants; unit: Participants] | 2
No stem cell transplant received [Count of Participants; unit: Participants] | 39
Oral posaconazole [Count of Participants; unit: Participants] | 59
Intravenous and oral posaconazole [Count of Participants; unit: Participants] | 5
Daily dose of posaconazole (mg/kg) [Median (Inter-Quartile Range); unit: mg/kg] | 4.5 [3.4 to 4.8]
Both stem cell transplantations received [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: C Reactive Protein Levels in mg/L (CRP) on Posaconazole Concentrations in mg/L
Description: Posaconazole drug exposure during treatment in different stages of inflammation. To determine the differences in concentrations between patients a random additive effect was used. Additionally, to correct for differences in intervals between observations a first-order autoregressive correlation was used. The Wald type III test was used to assess the influence of inflammation on posaconazole concentration.
Time Frame: 6 months after start of treatment
Measure: Median (Inter-Quartile Range); unit: mg/L
Groups:
- Posaconazole: Patients who received posaconazole for routine care
Arm/Group | Posaconazole
Number analyzed (Participants) | 64
mg/L
  Posaconazole concentration | 1.8 [1 to 2.9]
  C reactive protein | 23.5 [5 to 75]
Statistical Analysis 1: Comparison: Posaconazole; Test type: Other; p = 0.77, The Wald Type III test

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were evaluated from the start of the treatment up to 1 year.
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Groups:
- Posaconazole: Route of administration:
  Oral (MDR tablet), intravenous (infusion) Daily dose (mg/kg body weight): 3.75 (3.4-4.9)
Arm/Group | Posaconazole
All-Cause Mortality (participants affected / at risk) | 5/64
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 3/64
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=64)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) — Thrombocytes and leukocytes levels decreased after starting posaconazole, however another drug could have also caused that adverse event (cotrimoxazole).
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) — Patient had hypernatremia after starting posaconazole, calcium and potassium were normal and another alternative cause was diagnosed diabetes insipidus.
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1) — After starting posaconazole there was a slight increase in liver enzymes (ALAT, ASAT).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT02492802/Prot_SAP_000.pdf